CLINICAL TRIAL: NCT03981978
Title: Validity of Physical Activity Questionnaires in Persons Pursuing Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0398-19-EP
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Bariatric Surgery Candidate; Obesity
Keywords: physical activity; accelerometer; bariatric surgery; obesity
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Physical Activity — Self-report questionnaires assessing physical activity level.
  Other Names: Human Activity Profile Questionnaire; Godin-Shephard Leisure Time Physical Activity Questionnaire

SUMMARY:
The purpose of this study is to determine the validity of the Human Activity Profile and Godin self-report questionnaires of physical activity in persons seeking metabolic surgery.

DETAILED DESCRIPTION:
This cross-sectional study will collect subject's medical history, anthropometric measurements, physical activity data through an accelerometer worn on the wrist and indirect physical activity measures via the Human Activity Profile and Godin self-report questionnaires. We will collect clinical information from the medical record including predictors of physical activity level in obesity such as nutritional lab and co-morbid conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age >19
* BMI > 30
* Able to speak and understand English
* Consent to provide access to medical records for medical history
* Will receive weight loss procedure (sleeve gastrectomy or gastric bypass) at Nebraska Medicine
* Consent to wear an activity tracker device for 7 days after designated visits.

Exclusion Criteria:

• Age < 19

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients seeking bariatric surgery at University of Nebraska Medical Center/Nebraska Medicine
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Human Activity Profile Questionnaire | Baseline - Single time point
  Self-report questionnaire - indirect measure of physical activity

SECONDARY OUTCOMES:
Godin-Shephard Leisure Time Physical Activity (Godin) questionnaire | Baseline - Single time point
  Self-report questionnaire - indirect measure of physical activity
Accelerometer | Baseline - Single time point
  Direct measure of physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Laura D Bilek, PhD, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - University of Nebraska Medical Center, Bariatric Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Physical Activity Lab, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No